CLINICAL TRIAL: NCT07195357
Title: Erosive Tooth Wear, Dentin Hypersensitivity and Associated Risk Factors: An Observational, Cross-Sectional, Multi-Site, Epidemiological Study in the U.S." IU IRB# 28041
Brief Title: Multi-site Study to Look at Tooth Wear and Tooth Sensitivity and the Risk Factors Associated.
Status: Not yet recruiting | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: HALEON (Industry)
Responsible Party: Principal Investigator, Anderson T. Hara, DDS, MS, Indiana University
Other Study IDs: 28041
Record Dates: First submitted 2025-09-11; First posted 2025-09-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Dentin Hypersensitivity; Erosive Tooth Wear
Keywords: erosive tooth wear; ETW; Dentin hypersensitivity; DH; Tooth Sensitivity; Dental Erosion
MeSH Terms: conditions — Dentin Sensitivity; Tooth Erosion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults age 18 living in five different areas of the United States: The five areas are Indiana, Florida, California, Texas and North Carolina
  Interventions: Other: epidemiological

INTERVENTIONS:
Other: epidemiological — collection of data from all participating subjects involving tooth erosion examinations, tooth sensitivity and questionnaire data collection

SUMMARY:
The goal of this observational study is to learn about tooth wear and tooth sensistivity and reasons for these conditions in five locations throughout the United States. The main question it aims to answer is:

The main objective of this study is to determine tooth wear and tooth sensitivity in adults in the U.S., and to investigate their association with risk factors

DETAILED DESCRIPTION:
The primary goal of this observational, cross-sectional, multi-site epidemiological study is to determine the prevalence of erosive tooth wear (ETW) and dentin hypersensitivity (DH) in healthy adults of different age brackets in the U.S., and to investigate their association with risk factors. A secondary goal is to assess gingival recession (GR) and presence of non-carious cervical lesion (NCCL). A tertiary goal is to compare the U.S. data with those from previous studies conducted in Europe and China.

Study participants will be healthy dentate adults aged 18 or older, recruited from clinics in dental schools (study sites), located in the U.S. Up to 5 study sites geographically distributed in the five U.S. regions (Midwest, Northeast, Southeast, Southwest, West) will participate in the study, with the goal of enrolling approximately 500 participants per site (total n = 2500), distributed nearly equally across age brackets (18-27, 28-37, 38-47, 48-57, 58+), and between males and females. In each site, a study team will be assigned with at least an investigator dental practitioner (dentist or dental hygienist) and a study coordinator will be assigned for the recruitment, consenting, examination, and intraoral scanning of participants. The main site under the direction of the PI will also include a project manager and an examiner for the digital images. Each site will file the study protocol, consent and associated documents through their own IRB using the respective documents approved by the Indiana University IRB. Each site may make modifications to the documents as required per each site's IRB.

Consented participants that agree to take part on the study and that meet the study inclusion and exclusion criteria will have clinical and self-reported data collected in a single study visit. Data sources will include questionnaire on demographics and associated factors, standardized intra-oral scanning of the full mouth and video recording of participants reactions while submitted to a DH test. The 3D digital images obtained from the intra-oral scans will be used for the digital assessment of ETW using the BEWE index. Video recordings will be used for the scoring of DH using the Schiff index and self-reported assessments. All digital scans and video recordings collected from the study sites will be managed by the lead site (Oral Health Research Institute - OHRI) and BEWE, GR and NCCL assessments will be performed digitally by previously trained examiner(s).

Preliminary, descriptive level analyses will be performed for the questionnaire variables. For each scoring variable, frequency distributions will be produced and summarized showing the variation between different areas of the mouth. The main analyses will be at the patient level, and the relationship between patient-level measures of each explanatory variable will be examined by crosstabulations and regression analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 18 or over, of either gender.
2. Be attending a regularly scheduled appointment at the dental school.
3. Provide voluntary, written informed consent.
4. Understand and be willing, able and likely to comply with all study procedures and restrictions.
5. Be in good health (see exclusion criteria below).
6. Have a minimum of 10 teeth not including implants or teeth with crowns or bridges.

Exclusion Criteria:

1. Have any medical condition that could be expected to interfere with the subject's safety during the study period (including temporomandibular disorders).
2. Be incapable of responding to the questions.
3. Be an employee or a family relative of an employee of the sponsor.
4. Be using maxillary or mandibular orthodontic appliances, except lingual bar.
5. Have used analgesic (pain relieving) drugs or have used a topical analgesic in the preceding 12 h

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be idenified from five regions in the United states who meet the inclusion/exclusion criteria listed in this application
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence and severity of erosive tooth wear (ETW), assessed using the basic erosive wear examination (BEWE) index. | Five minute examination period
  ETW will be assessed on captured intraoral scans, for each tooth/subject using BEWE index. It will be performed by a previously trained and calibrated examiner. The BEWE scale presents 4 levels, from 0: no ETW to 3: most severe ETW.
Prevalence and severity of dentin hypersensitivity (DH) using the Schiff Sensitivity Index. | Five minute examination period
  DH will be assessed on recorded video files by a previously trained examiner, who will watch the videos and provide a Schiff score for each tooth/subject. The Schiff scale has 5 severity levels, ranging from 0: no DH to 4: severe DH.
Risk factors potentially associated to erosive tooth wear (ETW) and dentin hypersensitivity (DH), collected by questionnaires. | Ten minutes assessment period.
  Demographics and potential risk factors associated with ETW and DH will be collected from each subject by questionnaires. They will include:
  1. Demographic data; age, gender, socioeconomic status, education level achieved, location, race/ethnicity.
  2. Data on the participant's oral hygiene practices.
  3. Data about the participant's dentin hypersensitivity quality of life experience.
  4. Data on the participant's perception of their general oral health, toothwear and gum health.
  5. Data on the participant's perception of DH: intensity, duration, origin.
  6. Data on the evaluation of risk factors associated with ETW and DH.

SECONDARY OUTCOMES:
Gum tissue recession presence, assessed on captured intraoral scans by a trained examiner. | Five minute examination period
  A secondary outcome is presence (yes or no) of gum tissue recession (wearing away of the gum at the gumline), assessed by a trained examiner.

OTHER OUTCOMES:
Compare study data to previously collected data | 0
  ETW and DH prevalence and risk factors observed in this study (U.S. data) will be compared to those collected in previous studies similarly designed and conducted in Europe and China.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Dentistry -Oral Health Research Institute, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No